CLINICAL TRIAL: NCT06799754
Title: Evaluation Of The Change In Ovarian Reserve Following Medical Therapy In Patients With Endometriosis
Brief Title: Ovarian Reserve Following Medical Therapy in Patients With Endometriosis
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: EndoAMH
Record Dates: First submitted 2024-12-03; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-11

CONDITIONS: Endometriosis
Keywords: endometriosis; medical therapy; ovarian reserve
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to investigate whether there is an effect on ovarian reserve from medical therapy for endometriosis.

Although the therapeutic efficacy of medical hormone therapy on ovarian endometriosis has been proven in many scientific studies, none of these has shown an effect on ovarian reserve.

The aim of this study is to investigate whether there is a difference in ovarian reserve as measured by biochemical and ultrasound parameters before and after therapy.

DETAILED DESCRIPTION:
Endometriosis is a benign, chronic and recurrent condition characterised by the presence of endometrial glands and stroma outside the uterine cavity. Endometriosis is most frequently localised to the ovary (17 - 44%) and is found in 5-10% of women of childbearing age. In this group of patients, quantification of the ovarian reserve by means of serological and ultrasound markers, in particular antral follicular count (AFC) and blood levels of antimullerian hormone (AMH), is essential. Recent evidence shows that medical hormone therapy, currently the first choice of treatment, affects ovarian endometriosis in terms of volumetric reduction of endometriomas and reduction of local inflammation, but little is known about its effect on ovarian reserve.

Our study therefore aims to evaluate ovarian reserve in terms of AMH and AFC in patients with ovarian endometriosis treated with medical hormone therapy after discontinuation of the latter.

In the clinical trial, patients diagnosed with ovarian endometriosis with an indication for medical therapy undergo 3 blood samples for the determination of antimullerian hormone (AMH) at the same time as 3 medical examinations as per normal care procedure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and ultrasound diagnosis of ovarian endometriosis without indication for surgery
* Age between 18 and 40 years
* Patients desiring pregnancy
* Informed consent obtained

Exclusion Criteria:

* Endocrinological disorders (including thyroid dysfunction, hyperprolactinaemia and Cushing's syndrome)
* Previous ovarian surgery
* Suspected cyst malignancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with ovarian endometriosis desiring pregnancy with or without concomitant deep endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-07-19 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve in patients with ovarian endometriosis | Through study completion, an average of 4 years
  Evaluate the ovarian reserve at ultrasound and biochemical level in patients with ovarian endometriosis treated with medical therapy

SECONDARY OUTCOMES:
Follicle stimulating hormone (FSH) | Through study completion, an average of 4 years
  Quantification of follicle stimulating hormone (FSH) levels
Ultrasound assessment of ovarian volume and endometriosis cyst volume | Through study completion, an average of 4 years
  Ultrasound assessment of ovarian volume and endometriosis cyst volume
Ovarian reserve in patients with concomitant deep endometriosis compared to those with ovarian endometriosis alone | Through study completion, an average of 4 years
  Evaluation of a possible difference in ovarian reserve in patients with concomitant deep endometriosis compared to those with ovarian endometriosis alone

CONTACTS AND LOCATIONS:
Overall Officials: Renato Seracchioli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy